CLINICAL TRIAL: NCT03891524
Title: A Randomized, Open-Label, Study Drug-Dose Blind, Multicenter Study to Evaluate the Efficacy and Safety of JNJ-70033093 (BMS-986177), an Oral Factor XIa Inhibitor, Versus Subcutaneous Enoxaparin in Subjects Undergoing Elective Total Knee Replacement Surgery
Brief Title: A Study of JNJ-70033093 (BMS-986177) Versus Subcutaneous Enoxaparin in Participants Undergoing Elective Total Knee Replacement Surgery
Acronym: AXIOMATIC-TKR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CR108600; 70033093THR2001 (Other: Janssen Research & Development, LLC); 2018-004237-32 (EudraCT Number)
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Results first posted 2022-07-15 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Arthroplasty, Replacement, Knee
MeSH Terms: interventions — milvexian; Enoxaparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Treatment arms and study drug dose regimens will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- Group A: JNJ-70033093 25 mg + Placebo BID (Experimental): Participants will receive JNJ-70033093 25 milligram (mg) (1*25 mg capsule) and 1 placebo capsule twice daily (BID), orally for 10 to 14 postoperative days.
  Interventions: Drug: JNJ-70033093 25 mg; Drug: Placebo
- Group B: JNJ-70033093 50 mg BID (Experimental): Participants will receive JNJ-70033093 50 mg (2*25 mg capsules) BID orally for 10 to 14 postoperative days.
  Interventions: Drug: JNJ-70033093 50 mg
- Group C: JNJ-70033093 100 mg + Placebo BID (Experimental): Participants will receive JNJ-70033093 100 mg (1*100 mg capsule) and 1 placebo capsule BID orally for 10 to 14 postoperative days.
  Interventions: Drug: JNJ-70033093 100 mg; Drug: Placebo
- Group D: JNJ-70033093 200 mg BID (Experimental): Participants will receive JNJ-70033093 200 mg (2*100 mg capsules) BID orally for 10 to 14 postoperative days.
  Interventions: Drug: JNJ-70033093 200 mg
- Group E: JNJ-70033093 25 mg Once Daily + Placebo (Experimental): Participants will receive JNJ-70033093 25 mg (1*25 mg capsule) once daily and 1 placebo capsule in the morning and 2 placebo capsules in the evening, orally for 10 to 14 postoperative days.
  Interventions: Drug: JNJ-70033093 25 mg; Drug: Placebo
- Group F: JNJ-70033093 200 mg Once Daily + Placebo (Experimental): Participants will receive JNJ-70033093 200 mg (2*100 mg capsules in the morning) once daily and 2 placebo capsules in the evening, orally for 10 to 14 postoperative days.
  Interventions: Drug: JNJ-70033093 200 mg; Drug: Placebo
- Group G: JNJ-70033093 50 mg once daily + Placebo (Experimental): Participants will receive JNJ-70033093 50 mg (2*25 mg capsules in the morning) once daily and 2 placebo capsules in the evening, orally for 10 to 14 postoperative days.
  Interventions: Drug: JNJ-70033093 50 mg; Drug: Placebo
- Group I: Enoxaparin 40 mg Once Daily (Active Comparator): Participants will receive enoxaparin 40 mg once daily subcutaneously for 10 to 14 postoperative days.
  Interventions: Drug: Enoxaparin 40 mg

INTERVENTIONS:
Drug: JNJ-70033093 25 mg — Participants will receive JNJ-70033093 25 mg (1*25 mg capsule) BID (in Group A) or once daily (in Group E), orally for 10 to 14 postoperative days.
  Other Names: BMS-986177
  Arms: Group A: JNJ-70033093 25 mg + Placebo BID; Group E: JNJ-70033093 25 mg Once Daily + Placebo
Drug: JNJ-70033093 50 mg — Participants will receive JNJ-70033093 50 mg (2*25 mg capsules) BID orally for 10 to 14 postoperative days.
  Other Names: BMS-986177
  Arms: Group B: JNJ-70033093 50 mg BID; Group G: JNJ-70033093 50 mg once daily + Placebo
Drug: JNJ-70033093 100 mg — Participants will receive JNJ-70033093 100 mg (1*100 mg capsule) BID, orally for 10 to 14 postoperative days.
  Other Names: BMS-986177
  Arms: Group C: JNJ-70033093 100 mg + Placebo BID
Drug: JNJ-70033093 200 mg — Participants will receive JNJ-70033093 200 mg (2*100 mg capsules) BID (in Group D) or once daily (in Group F), orally for 10 to 14 postoperative days.
  Other Names: BMS-986177
  Arms: Group D: JNJ-70033093 200 mg BID; Group F: JNJ-70033093 200 mg Once Daily + Placebo
Drug: Placebo — Participants will receive placebo matching to JNJ-70033093, orally.
  Arms: Group A: JNJ-70033093 25 mg + Placebo BID; Group C: JNJ-70033093 100 mg + Placebo BID; Group E: JNJ-70033093 25 mg Once Daily + Placebo; Group F: JNJ-70033093 200 mg Once Daily + Placebo; Group G: JNJ-70033093 50 mg once daily + Placebo
Drug: Enoxaparin 40 mg — Participants will receive enoxaparin 40 mg once daily subcutaneously for 10 to 14 postoperative days.
  Arms: Group I: Enoxaparin 40 mg Once Daily

SUMMARY:
The purpose of this study is to determine the efficacy of JNJ-70033093 in preventing total venous thromboembolism (VTE) events (proximal and/or distal deep vein thrombosis [DVT] [asymptomatic confirmed by venography assessment or objectively confirmed symptomatic], nonfatal pulmonary embolism [PE], or any death) during the treatment period.

DETAILED DESCRIPTION:
JNJ-70033093 is an oral anticoagulant for prevention and treatment of thromboembolic events (for example, VTE) that binds and inhibits activated form of human coagulation Factor XI (FXIa) with high affinity and selectivity. The study will consist of 3 phases: up to 30-day screening phase before total knee replacement (TKR) surgery, 10 to14 day postoperative dosing phase, and 4-week follow-up phase. The hypothesis of this study is JNJ-70033093 reduces risk of total VTE during treatment period. The total duration of participation following randomization will be approximately 6 weeks. Efficacy evaluations include unilateral venography assessment of operated leg and assessments of symptomatic DVT, PE, or death. Safety evaluation includes adverse events, clinical laboratory tests, and physical examinations. The safety and efficacy will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable and appropriate for anticoagulant prophylaxis as determined by the investigator on the basis of physical examination, medical history, and vital signs performed as part of screening for elective total knee replacement (TKR) surgery
* Medically stable and appropriate for anticoagulant prophylaxis on the basis of clinical laboratory tests performed as part of local standard-of-care as part of screening for elective TKR surgery
* Has plans to undergo an elective primary unilateral TKR surgery
* A woman must be- a) Not of childbearing potential; b) Of childbearing potential and practicing a highly effective method of contraception (failure rate of less than [<]1 percent [%] per year when used consistently and correctly) and agrees to remain on a highly effective method for the duration of study drug with JNJ-70033093 plus 5 half-lives of study drug plus 30 days (duration of ovulatory cycle) for a total of 34 days after the completion of treatment, pregnancy testing (serum or urine) prior to the first dose of study drug
* Willing and able to adhere to the lifestyle restrictions specified in this protocol

Exclusion Criteria:

* History of any condition for which the use of low molecular-weight heparin (LMWH) is not recommended in the opinion of the investigator (for example, previous allergic reaction, creatinine clearance <30 milliliter per minute [mL/minute])
* History of severe hepatic impairment
* Planned bilateral revision or unicompartmental procedure
* Unable to undergo venography (for example, due to contrast agent allergy, poor venous access, or impaired renal function that would increase the risk of contrast-induced nephropathy
* Known previous pulmonary embolism (PE) or deep vein thrombosis (DVT) in either lower extremity

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1242 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (117):
- United States (9):
  - Central Research Associates, Inc., Birmingham, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - Bowen Hefley Orthopedics, Little Rock, Arkansas
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Denver Metro Orthopedics, PC, Englewood, Colorado
  - DMI Research, Pinellas Park, Florida
  - Gulfcoast Research Institute, Sarasota, Florida
  - University Orthopedic and Joint Replacement Center, Tamarac, Florida
  - Memorial Hermann Memorial City Medical Center, Houston, Texas
- Argentina (7):
  - Hospital Britanico de Buenos Aires, Buenos Aires
  - Clinica Adventista Belgrano, CABA
  - Hospital San Roque, Córdoba
  - Clínica Chutro, Córdoba
  - Hospital Italiano La Plata, La Plata
  - Instituto de Investigaciones Clinicas Rosario, Rosario
  - Sanatorio Corporación Médica de General San Martín, San Martín
- Belgium (4):
  - ZNA Middelheim, Antwerp
  - Ziekenhuis Oost-Limburg, Genk
  - Jessa Ziekenhuis, Hasselt
  - ZNA Jan Palfijn, Merksem
- Brazil (3):
  - Hospital Sao Francisco de Assis, Belo Horizonte
  - Hospital e Maternidade Dr Christovao da Gama S.A, Santo André
  - Hospital Estadual Mario covas, Santo André
- Bulgaria (5):
  - University Multiprofile Hospital for Active Treatment Dr. Georgi Stranski, Pleven
  - Acibadem City Clinic Tokuda Hospital, Sofa
  - University Multiprofile Hospital Sofiamed Sofia, Sofia
  - MHAT Tzaritza Joanna, Sofia
  - Medical Center - Medical Complex BEROE EOOD, Stara Zagora
- Canada (4):
  - Lakeridge Health, Ajax, Ontario
  - Hamilton Health Sciences Corporation, Hamilton, Ontario
  - The Ottawa Hospital Research Institute, Ottawa, Ontario
  - Medical Investigative and Clinical Evaluation Inc, Windsor, Ontario
- Greece (4):
  - General Hospital of Attiki 'KAT', Kifissia
  - General Hospital of Nea Ionia 'Konstantopoulio', Nea Ionia
  - University General Hospital of Rio Patras, Pátrai
  - Papageorgiou General Hospital, Thessaloniki
- Hungary (8):
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem, Debrecen
  - Petz Aladar Megyei Oktato Korhaz, Gyõr
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Bacs-kiskun Megyei Korhaz, Kecskemét
  - Szegedi Tudomanyegyetem, Szeged
  - Fejer Varmegyei Szent Gyorgy Egyetemi Oktatokorhaz, Székesfehérvár
  - MAV Korhaz es Rendelointezet, Szolnok
- Israel (4):
  - Rambam Medical Center, Haifa
  - Carmel Medical Center, Haifa
  - Meir Medical Center, Kfar Saba
  - Kaplan Medical Center, Rehovot
- Italy (6):
  - Cliniche Humanitas Gavazzeni, Bergamo
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Istituto Ortopedico Rizzoli, Bologna
  - Policlinico S. Matteo, Pavia
  - Istituto Clinico Humanitas, Rozzano
  - A.O.U. Città della Salute e della Scienza, Torino
- Japan (15):
  - Matsudo City General Hospital, Chiba
  - Hakodate Goryoukaku Hospital, Hakodate
  - Japanese Red Cross Hamamatsu Hospital, Hamamatsu
  - Itami City Hospital, Itami-shi
  - Yonemori Hospital, Kagoshima
  - Japan Community Health care Organization Kyushu Hospital, Kitakyushu-shi
  - Marunouchi Hospital, Matsumoto
  - Chubu Rosai Hospital, Nagoya
  - Juntendo University Nerima Hospital, Nerima-Ku
  - National Hospital Organization Okayama Medical Center, Okayama
  - Yuuai Medical Center, Okinawa
  - Japan Community Health Care Organization Saitama Medical Center, Saitama
  - Saitama City Hospital, Saitama-shi
  - Nagano Prefectural Shinshu Medical Center, Suzaka
  - Juntendo University Hospital, Tokyo
- Poland (9):
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej w Bielsku Podlaskim Oddzial Urazowo Ortopedyczny, Bielsk Podlaski
  - Szpital Ogolny im. W. Ginela, Oddzial Urazowo-Ortopedyczny, Grajewo
  - Wojewodzki Szpital Zespolony w Kielcach, Klinika Chirurgii Ortopedyczno-Urazowej, Kielce
  - Oddzial Ortopedii i Traumatologii Narzadu Ruchu Szpital Specjalistyczny im Ludwika Rydygiera, Krakow
  - CSK UM Klinika Ortopedii, Lodz
  - Oddzial Urazowo-Ortopedyczny Wojewodzki Szpital Specjalistyczny, Lublin
  - Oddzial Ortopedii Specjalistyczny Szpital im. E.Szczeklika, Tarnów
  - Oddzial Chirurgii Urazowej iOrtopedycznej Wojewodzki Szpital Brodnowski SPZOZ, Warsaw
  - Uniwersytecki Szpital Kliniczny im Jana Mikulicza Radeckiego we Wroclawiu, Wroclaw
- Portugal (5):
  - Centro Hospitalar do Baixo Vouga - Hospital Infante Dom Pedro, Aveiro
  - Hosp de Cascais, Cascais
  - H. Santo António - Centro Hospitalar do Porto, Porto
  - CHS - Hosp. Orto. Sant'Iago do Outao, Setúbal
  - ULSAM, EPE - Hospital de Santa Luzia, Viana do Castelo
- Russia (7):
  - National Medical Research Center of Traumatology and Orthopaedics n.a. G.A. Ilizarov, Kurgan
  - Private Healthcare Institution 'Clinical Hospital 'RZD-Medcine' n.a. N.A.Semashko', Moscow
  - Privolzhsky Regional Medical Center of Federal Medical and Biological Agency, Nizhny Novgorod
  - National medical research center of Traumatology and Orthopaedics n.a. R.R.Vreden, Saint Petersburg
  - State Healthcare Institution Samara Regional Clinical Hospital named after V.D.Seredavin, Samara
  - Smolensk Federal Center of Traumatology, Orthopedics and Endoprothesis Replacement, Smolensk
  - Sochi City Hospital #4, Sochi
- South Africa (2):
  - Steve Biko Academic Hospital, Pretoria
  - Clinical Project Research SA, Worcester
- Spain (11):
  - Hosp. Univ. Fundacion Alcorcon, Alcorcón
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Univ. de Bellvitge, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Complejo Hospitalario de Jaen, Jaén
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Corporacio Sanitari Parc Tauli, Sabadell
  - Hosp. Clinico Univ. de Valencia, Valencia
  - Hosp. Univ. I Politecni La Fe, Valencia
- Turkey (Türkiye) (7):
  - Adana City Hospital, Adana
  - Diskapi Yildırim Beyazid Training and Research Hospital, Ankara
  - Yıldırım Beyazıt University Yenimahalle Training and Research Hospital, Ankara
  - Antalya Training And Research Hospital, Antalya
  - Bakirkoy Training and Research Hospital, Istanbul
  - Sisli Etfal Research Training Hospital, Istanbul
  - Izmir Tepecik Training and Research Hospital, Izmir
- Ukraine (7):
  - Ivano-Frankivsk Regional Clinical Hospital, Ivano-Frankivsk
  - Institute of Spine and JointPathology named after Prof.Sytenko of NationalAcademy of MedicalSciences, Kharkiv
  - Municipal Institution of Health Care 'Kharkiv Regional Clinical Traumatology Hospital', Kharkiv
  - Kyiv Regional Clinical Hospital, Kyiv
  - Communal Institution of Lviv Regional Council 'Lypa Lviv Regional Hospital', Lviv-Vynnyky
  - Municipal Non-profit Enterprise 'Odesa Regional Clinical Hospital' Odesa Regional Council, Odesa
  - Vinnytsya Regional Clinical Hospital named after M.I.Pirogov, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinicaltrials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Whiteson HZ, Frishman WH. Factor XI/XIa Inhibitors: A New Approach to Anticoagulation. Cardiol Rev. 2025 Jul-Aug 01;33(4):306-311. doi: 10.1097/CRD.0000000000000624. Epub 2023 Dec 1. PMID 38038437
- [Derived] Weitz JI, Strony J, Ageno W, Gailani D, Hylek EM, Lassen MR, Mahaffey KW, Notani RS, Roberts R, Segers A, Raskob GE; AXIOMATIC-TKR Investigators. Milvexian for the Prevention of Venous Thromboembolism. N Engl J Med. 2021 Dec 2;385(23):2161-2172. doi: 10.1056/NEJMoa2113194. Epub 2021 Nov 15. PMID 34780683

RESULTS

PARTICIPANT FLOW:
Groups:
- JNJ-70033093 25 mg Once Daily + Placebo: Participants received JNJ-70033093 25 milligrams (mg) (1*25 mg capsule) once daily and 1 placebo capsule in the morning and 2 placebo capsules in the evening, orally for 10 to 14 postoperative days.
- JNJ-70033093 50 mg Once Daily + Placebo: Participants received JNJ-70033093 50 mg (2*25 mg capsules in the morning) once daily and 2 placebo capsules in the evening, orally for 10 to 14 postoperative days.
- JNJ-70033093 25 mg + Placebo Twice Daily (BID): Participants received JNJ-70033093 25 mg (1*25 mg capsule) and 1 placebo capsule twice daily (BID), orally for 10 to 14 postoperative days.
- JNJ-70033093 50 mg BID: Participants received JNJ-70033093 50 mg (2*25 mg capsules) BID orally for 10 to 14 postoperative days.
- JNJ-70033093 200 mg Once Daily + Placebo: Participants received JNJ-70033093 200 mg (2*100 mg capsules in the morning) once daily and 2 placebo capsules in the evening, orally for 10 to 14 postoperative days.
- JNJ-70033093 100 mg + Placebo BID: Participants received JNJ-70033093 100 mg (1*100 mg capsule) and 1 placebo capsule BID orally for 10 to 14 postoperative days.
- JNJ-70033093 200 mg BID: Participants received JNJ-70033093 200 mg (2*100 mg capsules) BID orally for 10 to 14 postoperative days.
- Enoxaparin 40 mg Once Daily: Participants received enoxaparin 40 mg once daily subcutaneously for 10 to 14 postoperative days.
Period: Overall Study
Arm/Group | JNJ-70033093 25 mg Once Daily + Placebo | JNJ-70033093 50 mg Once Daily + Placebo | JNJ-70033093 25 mg + Placebo Twice Daily (BID) | JNJ-70033093 50 mg BID | JNJ-70033093 200 mg Once Daily + Placebo | JNJ-70033093 100 mg + Placebo BID | JNJ-70033093 200 mg BID | Enoxaparin 40 mg Once Daily
Started | 34 | 150 | 153 | 150 | 149 | 152 | 153 | 301
Safety Analysis Set | 33 | 150 | 148 | 148 | 147 | 149 | 148 | 296
Completed | 34 | 149 | 151 | 149 | 147 | 150 | 151 | 299
Not Completed | 0 | 1 | 2 | 1 | 2 | 2 | 2 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 1 | 2 | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | JNJ-70033093 25 mg Once Daily + Placebo | JNJ-70033093 50 mg Once Daily + Placebo | JNJ-70033093 25 mg + Placebo Twice Daily (BID) | JNJ-70033093 50 mg BID | JNJ-70033093 200 mg Once Daily + Placebo | JNJ-70033093 100 mg + Placebo BID | JNJ-70033093 200 mg BID | Enoxaparin 40 mg Once Daily | Total
Number analyzed (Participants) | 34 | 150 | 153 | 150 | 149 | 152 | 153 | 301 | 1242
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (5.74) | 67.9 (8.03) | 68.4 (8.49) | 68.8 (8.17) | 68 (8.25) | 67 (8) | 68.6 (7.76) | 67.8 (7.97) | 68 (8.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 107 | 113 | 108 | 108 | 102 | 106 | 208 | 876
  Male | 10 | 43 | 40 | 42 | 41 | 50 | 47 | 93 | 366
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 21 | 19 | 20 | 20 | 14 | 14 | 42 | 156
  Not Hispanic or Latino | 28 | 121 | 126 | 125 | 125 | 129 | 133 | 250 | 1037
  Unknown or Not Reported | 0 | 8 | 8 | 5 | 4 | 9 | 6 | 9 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
  Asian | 0 | 22 | 17 | 16 | 17 | 16 | 16 | 32 | 136
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 4
  Black or African American | 0 | 1 | 2 | 1 | 0 | 3 | 1 | 4 | 12
  White | 34 | 124 | 134 | 132 | 129 | 132 | 136 | 260 | 1081
  More than one race | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 2 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  Asia | 0 | 22 | 16 | 16 | 16 | 16 | 16 | 32 | 134
  Europe | 21 | 55 | 65 | 65 | 64 | 64 | 65 | 129 | 528
  South America | 0 | 9 | 7 | 6 | 7 | 7 | 6 | 13 | 55
  North America | 5 | 19 | 20 | 19 | 19 | 19 | 21 | 38 | 160
  Western Europe | 8 | 45 | 45 | 44 | 43 | 46 | 45 | 89 | 365

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Total Venous Thromboembolism (VTE) (CEC-adjudicated)
Description: Total VTE was defined as the composite of clinical events committee (CEC)-adjudicated proximal and/or distal Deep Vein Thrombosis (DVT) (asymptomatic confirmed by venography assessment of the operated leg or objectively confirmed symptomatic), nonfatal pulmonary embolism (PE), or any death.
Time Frame: Up to Day 14
Population: The modified Intent-to-treat (mITT) analysis set included all intent-to-treat (ITT) participants who received at least 1 dose of study drug with an evaluable venography assessment or a confirmed symptomatic proximal DVT, PE or death as adjudicated by the CEC.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-70033093 25 mg Once Daily + Placebo | JNJ-70033093 50 mg Once Daily + Placebo | JNJ-70033093 25 mg + Placebo Twice Daily (BID) | JNJ-70033093 50 mg BID | JNJ-70033093 200 mg Once Daily + Placebo | JNJ-70033093 100 mg + Placebo BID | JNJ-70033093 200 mg BID | Enoxaparin 40 mg Once Daily
Number analyzed (Participants) | 28 | 127 | 129 | 124 | 123 | 134 | 131 | 252
Participants | 7 | 30 | 27 | 14 | 8 | 12 | 10 | 54

2. Secondary Outcome: Number of Participants With Any Bleeding Event (CEC-adjudicated)
Description: Any bleeding was defined as the composite of major bleeding according to the International Society on Thrombosis and Haemostasis (ISTH) criteria modified for the surgical setting, clinically relevant nonmajor bleeding events, or minimal bleeding events as assessed by the CEC.
Time Frame: Up to Day 14; Up to Day 52
Population: The safety analysis set was a subset of the ITT analysis set, consisting of all ITT participants who received at least 1 dose (partial or complete) of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-70033093 25 mg Once Daily + Placebo | JNJ-70033093 50 mg Once Daily + Placebo | JNJ-70033093 25 mg + Placebo Twice Daily (BID) | JNJ-70033093 50 mg BID | JNJ-70033093 200 mg Once Daily + Placebo | JNJ-70033093 100 mg + Placebo BID | JNJ-70033093 200 mg BID | Enoxaparin 40 mg Once Daily
Number analyzed (Participants) | 33 | 150 | 148 | 148 | 147 | 149 | 148 | 296
Participants
  Up to Day 14 | 0 | 8 | 2 | 7 | 11 | 7 | 6 | 12
  Up to Day 52 | 0 | 8 | 2 | 7 | 11 | 7 | 6 | 12

3. Secondary Outcome: Number of Participants With Total VTE (CEC-adjudicated)
Description: Total VTE was defined as the composite of (CEC-adjudicated) proximal and/or DVT (asymptomatic confirmed by venography assessment of the operated leg or objectively confirmed symptomatic), nonfatal PE, or any death.
Time Frame: Up to Day 52
Population: The mITT analysis set included all the participants in mITT at Day 14 plus the participants who had symptomatic/asymptomatic VTE events (DVT, non-fatal PE or any death) after day 17 through day 52. Also included the participants whose venography result was not evaluable distal but no proximal clot.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-70033093 25 mg Once Daily + Placebo | JNJ-70033093 50 mg Once Daily + Placebo | JNJ-70033093 25 mg + Placebo Twice Daily (BID) | JNJ-70033093 50 mg BID | JNJ-70033093 200 mg Once Daily + Placebo | JNJ-70033093 100 mg + Placebo BID | JNJ-70033093 200 mg BID | Enoxaparin 40 mg Once Daily
Number analyzed (Participants) | 28 | 128 | 129 | 124 | 123 | 135 | 131 | 253
Participants | 7 | 30 | 27 | 14 | 8 | 12 | 10 | 54

4. Secondary Outcome: Number of Participants With Composite of Major and Clinically Relevant Nonmajor Bleeding (CRNM) Events (CEC-adjudicated)
Description: Composite of Major bleeding event (BE): Fatal bleeding; bleeding that is symptomatic and occurs in critical area/organ and/or; extrasurgical site bleeding causing fall in Hemoglobin (Hb) level of 20 grams per liter (g/L) or more, or leading to transfusion of 2 or more units of whole blood or red cells with temporal association within 24-48 hours to bleeding, and/or; surgical site bleeding that requires second intervention open, arthroscopic, endovascular,or hemarthrosis resulting in prolonged hospitalization, deep wound infection and/or either unexpected and prolonged and/or sufficiently large to cause hemodynamic instability. CRNM bleeding: acute clinically overt bleeding that does not satisfy additional criteria required for bleeding event to be defined as major BE is still considered clinically relevant for example: Epistaxis, Gastrointestinal bleed,Hematuria,Bruising/ecchymosis,Hemoptysis,Hematoma.
Time Frame: Up to Day 14, Up to Day 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-70033093 25 mg Once Daily + Placebo | JNJ-70033093 50 mg Once Daily + Placebo | JNJ-70033093 25 mg + Placebo Twice Daily (BID) | JNJ-70033093 50 mg BID | JNJ-70033093 200 mg Once Daily + Placebo | JNJ-70033093 100 mg + Placebo BID | JNJ-70033093 200 mg BID | Enoxaparin 40 mg Once Daily
Number analyzed (Participants) | 33 | 150 | 148 | 148 | 147 | 149 | 148 | 296
Participants
  Up to Day 14 | 0 | 2 | 0 | 2 | 1 | 1 | 1 | 5
  Up to Day 52 | 0 | 2 | 0 | 2 | 2 | 1 | 1 | 5

5. Secondary Outcome: Number of Participants With Major Bleeding Events (CEC-adjudicated)
Description: Number of participants with major BE (adjudicated by CEC) were reported. Major Bleeding events were defined as: fatal bleeding; bleeding that is symptomatic and occurs in critical area/organ and/or; extrasurgical site bleeding causing fall in Hb level of 20 g/L or more, or leading to transfusion of 2 or more units of whole blood or red cells with temporal association within 24-48 hours to bleeding, and/or; requires second intervention open, arthroscopic, endovascular, or hemarthrosis resulting in prolonged hospitalization or a deep wound infection and/or; either unexpected and prolonged and/or sufficiently large to cause hemodynamic instability.
Time Frame: Up to Day 14; Up to Day 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-70033093 25 mg Once Daily + Placebo | JNJ-70033093 50 mg Once Daily + Placebo | JNJ-70033093 25 mg + Placebo Twice Daily (BID) | JNJ-70033093 50 mg BID | JNJ-70033093 200 mg Once Daily + Placebo | JNJ-70033093 100 mg + Placebo BID | JNJ-70033093 200 mg BID | Enoxaparin 40 mg Once Daily
Number analyzed (Participants) | 33 | 150 | 148 | 148 | 147 | 149 | 148 | 296
Participants
  Up to Day 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Up to Day 52 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

6. Secondary Outcome: Number of Participants With CRNM Bleeding Events (CEC-adjudicated)
Description: Number of participants with CRNM bleeding events (adjudicated by CEC) were reported. CRNM bleeding: acute clinically overt bleeding that does not satisfy additional criteria required for bleeding event to be defined as major BE is still considered clinically relevant for example: epistaxis, gastrointestinal bleed, hematuria, bruising/ecchymosis, hemoptysis, hematoma.
Time Frame: Up to Day 14; Up to Day 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-70033093 25 mg Once Daily + Placebo | JNJ-70033093 50 mg Once Daily + Placebo | JNJ-70033093 25 mg + Placebo Twice Daily (BID) | JNJ-70033093 50 mg BID | JNJ-70033093 200 mg Once Daily + Placebo | JNJ-70033093 100 mg + Placebo BID | JNJ-70033093 200 mg BID | Enoxaparin 40 mg Once Daily
Number analyzed (Participants) | 33 | 150 | 148 | 148 | 147 | 149 | 148 | 296
Participants
  Up to Day 14 | 0 | 2 | 0 | 2 | 1 | 1 | 1 | 4
  Up to Day 52 | 0 | 2 | 0 | 2 | 2 | 1 | 1 | 4

7. Secondary Outcome: Number of Participants With Minimal Bleeding Events (CEC-adjudicated)
Description: Number of participants with minimal bleeding events (adjudicated by CEC) were reported. Minimal bleeding event was defined as any bleeding event not met major or CRNM criteria. CRNM bleeding: acute clinically overt bleeding that does not satisfy additional criteria required for bleeding event to be defined as major BE is still considered clinically relevant for example: epistaxis, gastrointestinal bleed, hematuria, bruising/ecchymosis, hemoptysis, hematoma.
Time Frame: Up to Day 14; Up to Day 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-70033093 25 mg Once Daily + Placebo | JNJ-70033093 50 mg Once Daily + Placebo | JNJ-70033093 25 mg + Placebo Twice Daily (BID) | JNJ-70033093 50 mg BID | JNJ-70033093 200 mg Once Daily + Placebo | JNJ-70033093 100 mg + Placebo BID | JNJ-70033093 200 mg BID | Enoxaparin 40 mg Once Daily
Number analyzed (Participants) | 33 | 150 | 148 | 148 | 147 | 149 | 148 | 296
Participants
  Up to Day 14 | 0 | 6 | 2 | 5 | 8 | 7 | 4 | 8
  Up to Day 52 | 0 | 6 | 2 | 5 | 9 | 7 | 5 | 8

8. Secondary Outcome: Number of Participants With Major or CRNM Bleeding Events (CEC-adjudicated)
Description: Major Bleeding events were defined as: fatal bleeding; bleeding that is symptomatic and occurs in critical area/organ and/or; extrasurgical site bleeding causing fall in Hb level of 20 g/L or more, or leading to transfusion of 2 or more units of whole blood or red cells with temporal association within 24-48 hours to bleeding, and/or; requires second intervention open, arthroscopic, endovascular, or hemarthrosis resulting in prolonged hospitalization or a deep wound infection and/or; either unexpected and prolonged and/or sufficiently large to cause hemodynamic instability. CRNM bleeding: acute clinically overt bleeding that does not satisfy additional criteria required for bleeding event to be defined as major BE is still considered clinically relevant for example: epistaxis, gastrointestinal bleed, hematuria, bruising/ecchymosis, hemoptysis, hematoma.
Time Frame: Up to Day 14; Up to Day 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-70033093 25 mg Once Daily + Placebo | JNJ-70033093 50 mg Once Daily + Placebo | JNJ-70033093 25 mg + Placebo Twice Daily (BID) | JNJ-70033093 50 mg BID | JNJ-70033093 200 mg Once Daily + Placebo | JNJ-70033093 100 mg + Placebo BID | JNJ-70033093 200 mg BID | Enoxaparin 40 mg Once Daily
Number analyzed (Participants) | 33 | 150 | 148 | 148 | 147 | 149 | 148 | 296
Participants
  Up to Day 14 | 0 | 2 | 0 | 2 | 1 | 1 | 1 | 5
  Up to Day 52 | 0 | 2 | 0 | 2 | 2 | 1 | 1 | 5

9. Secondary Outcome: Number of Participants With Major VTE (CEC-adjudicated)
Description: Number of participants with major VTE (adjudicated by CEC) were reported. Major VTE was defined as a composite of proximal DVT (asymptomatic confirmed by venography or objectively confirmed symptomatic), nonfatal PE, or any death.
Time Frame: Up to Day 52
Population: The mITT analysis set included all the participants in mITT at Day 14 plus the participants who had symptomatic/asymptomatic VTE events (DVT, non-fatal PE or any death) after day 17 through day 52.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-70033093 25 mg Once Daily + Placebo | JNJ-70033093 50 mg Once Daily + Placebo | JNJ-70033093 25 mg + Placebo Twice Daily (BID) | JNJ-70033093 50 mg BID | JNJ-70033093 200 mg Once Daily + Placebo | JNJ-70033093 100 mg + Placebo BID | JNJ-70033093 200 mg BID | Enoxaparin 40 mg Once Daily
Number analyzed (Participants) | 28 | 128 | 129 | 124 | 123 | 135 | 131 | 253
Participants | 0 | 2 | 1 | 1 | 0 | 2 | 0 | 4

10. Secondary Outcome: Number of Participants With Major VTE (CEC-adjudicated)
Description: as for outcome 9
Time Frame: Up to Day 14
Population: The mITT analysis set at Day 14 included all ITT participants who received at least 1 dose of study drug with an evaluable venography assessment or a confirmed symptomatic VTE event (DVT, non-fatal PE or any death).
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-70033093 25 mg Once Daily + Placebo | JNJ-70033093 50 mg Once Daily + Placebo | JNJ-70033093 25 mg + Placebo Twice Daily (BID) | JNJ-70033093 50 mg BID | JNJ-70033093 200 mg Once Daily + Placebo | JNJ-70033093 100 mg + Placebo BID | JNJ-70033093 200 mg BID | Enoxaparin 40 mg Once Daily
Number analyzed (Participants) | 28 | 127 | 129 | 124 | 123 | 134 | 131 | 252
Participants | 0 | 2 | 1 | 1 | 0 | 2 | 0 | 4

11. Secondary Outcome: Number of Participants With Proximal Deep Vein Thrombosis (DVT) (CEC-adjudicated)
Description: Number of participants with proximal DVT (adjudicated by CEC) were reported. DVT asymptomatic confirmed by venography assessment of the operated leg or objectively confirmed symptomatic.
Time Frame: Up to Day 14
Population: The mITT analysis set at Day 14 includes all ITT participants who received at least 1 dose of study drug with an evaluable venography assessment or a confirmed symptomatic VTE event (DVT, non-fatal PE or any death). Also includes the subjects whose venography result is not evaluable distal but no proximal clot.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-70033093 25 mg Once Daily + Placebo | JNJ-70033093 50 mg Once Daily + Placebo | JNJ-70033093 25 mg + Placebo Twice Daily (BID) | JNJ-70033093 50 mg BID | JNJ-70033093 200 mg Once Daily + Placebo | JNJ-70033093 100 mg + Placebo BID | JNJ-70033093 200 mg BID | Enoxaparin 40 mg Once Daily
Number analyzed (Participants) | 29 | 134 | 133 | 128 | 128 | 136 | 135 | 259
Participants
  Asymptomatic | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Symptomatic | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Proximal DVT (CEC-adjudicated)
Description: Number of participants with proximal DVT (CEC-adjudicated) were reported. DVT asymptomatic confirmed by venography assessment of the operated leg or objectively confirmed symptomatic.
Time Frame: Up to Day 52
Population: The mITT analysis set included all the participants in mITT at Day 14 plus the participants who had symptomatic/asymptomatic VTE events (DVT, non-fatal PE or any death) after day 17 through day 52 and also included the participants whose venography result was not evaluable distal but no proximal clot.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-70033093 25 mg Once Daily + Placebo | JNJ-70033093 50 mg Once Daily + Placebo | JNJ-70033093 25 mg + Placebo Twice Daily (BID) | JNJ-70033093 50 mg BID | JNJ-70033093 200 mg Once Daily + Placebo | JNJ-70033093 100 mg + Placebo BID | JNJ-70033093 200 mg BID | Enoxaparin 40 mg Once Daily
Number analyzed (Participants) | 29 | 135 | 133 | 128 | 128 | 137 | 135 | 260
Participants
  Asymptomatic | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Symptomatic | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Distal DVT (CEC-adjudicated)
Description: Number of participants with distal DVT (CEC-adjudicated) were reported. DVT asymptomatic confirmed by venography assessment of the operated leg or objectively confirmed symptomatic.
Time Frame: Up to Day 14
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-70033093 25 mg Once Daily + Placebo | JNJ-70033093 50 mg Once Daily + Placebo | JNJ-70033093 25 mg + Placebo Twice Daily (BID) | JNJ-70033093 50 mg BID | JNJ-70033093 200 mg Once Daily + Placebo | JNJ-70033093 100 mg + Placebo BID | JNJ-70033093 200 mg BID | Enoxaparin 40 mg Once Daily
Number analyzed (Participants) | 28 | 127 | 129 | 124 | 123 | 134 | 131 | 252
Participants
  Asymptomatic | 7 | 27 | 26 | 13 | 8 | 10 | 10 | 50
  Symptomatic | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0

14. Secondary Outcome: Number of Participants With Distal DVT (CEC-adjudicated)
Description: Number of participants with distal DVT (adjudicated by CEC) were reported. DVT asymptomatic confirmed by venography assessment of the operated leg or objectively confirmed symptomatic.
Time Frame: Up to Day 52
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-70033093 25 mg Once Daily + Placebo | JNJ-70033093 50 mg Once Daily + Placebo | JNJ-70033093 25 mg + Placebo Twice Daily (BID) | JNJ-70033093 50 mg BID | JNJ-70033093 200 mg Once Daily + Placebo | JNJ-70033093 100 mg + Placebo BID | JNJ-70033093 200 mg BID | Enoxaparin 40 mg Once Daily
Number analyzed (Participants) | 28 | 128 | 129 | 124 | 123 | 135 | 131 | 253
Participants
  Asymptomatic | 7 | 27 | 26 | 13 | 8 | 10 | 10 | 50
  Symptomatic | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 0

15. Secondary Outcome: Number of Participants With Nonfatal Pulmonary Embolism (PE) (CEC-adjudicated)
Description: Number of participants with nonfatal PE (adjudicated by CEC) were reported.
Time Frame: Up to Day 14
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-70033093 25 mg Once Daily + Placebo | JNJ-70033093 50 mg Once Daily + Placebo | JNJ-70033093 25 mg + Placebo Twice Daily (BID) | JNJ-70033093 50 mg BID | JNJ-70033093 200 mg Once Daily + Placebo | JNJ-70033093 100 mg + Placebo BID | JNJ-70033093 200 mg BID | Enoxaparin 40 mg Once Daily
Number analyzed (Participants) | 28 | 127 | 129 | 124 | 123 | 134 | 131 | 252
Participants | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1

16. Secondary Outcome: Number of Participants With Nonfatal Pulmonary Embolism (PE) (CEC-adjudicated)
Description: Number of participants with nonfatal PE (adjudicated by CEC) were reported.
Time Frame: Up to Day 52
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-70033093 25 mg Once Daily + Placebo | JNJ-70033093 50 mg Once Daily + Placebo | JNJ-70033093 25 mg + Placebo Twice Daily (BID) | JNJ-70033093 50 mg BID | JNJ-70033093 200 mg Once Daily + Placebo | JNJ-70033093 100 mg + Placebo BID | JNJ-70033093 200 mg BID | Enoxaparin 40 mg Once Daily
Number analyzed (Participants) | 28 | 128 | 129 | 124 | 123 | 135 | 131 | 253
Participants | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1

17. Secondary Outcome: Number of Participants With Deaths (CEC-adjudicated)
Description: Number of participants with deaths (CEC-adjudicated) were reported.
Time Frame: Up to Day 14
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-70033093 25 mg Once Daily + Placebo | JNJ-70033093 50 mg Once Daily + Placebo | JNJ-70033093 25 mg + Placebo Twice Daily (BID) | JNJ-70033093 50 mg BID | JNJ-70033093 200 mg Once Daily + Placebo | JNJ-70033093 100 mg + Placebo BID | JNJ-70033093 200 mg BID | Enoxaparin 40 mg Once Daily
Number analyzed (Participants) | 28 | 127 | 129 | 124 | 123 | 134 | 131 | 252
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

18. Secondary Outcome: Number of Participants With Deaths (CEC-adjudicated)
Description: Number of participants with deaths (CEC-adjudicated) were reported.
Time Frame: Up to Day 52
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-70033093 25 mg Once Daily + Placebo | JNJ-70033093 50 mg Once Daily + Placebo | JNJ-70033093 25 mg + Placebo Twice Daily (BID) | JNJ-70033093 50 mg BID | JNJ-70033093 200 mg Once Daily + Placebo | JNJ-70033093 100 mg + Placebo BID | JNJ-70033093 200 mg BID | Enoxaparin 40 mg Once Daily
Number analyzed (Participants) | 28 | 128 | 129 | 124 | 123 | 135 | 131 | 253
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

19. Secondary Outcome: Apparent Clearance (CL/F) of JNJ-70033093
Description: Apparent clearance of a drug was defined as a measure of the rate at which a drug got metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed.
Time Frame: Up to Day 14
Population: The pharmacokinetic (PK) analysis set consisted of participants who received at least 1 dose of milvexian and had at least one valid blood sample drawn for PK analysis. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure. This outcome measure was planned to be analyzed for overall participants and not group wise.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/h)
Groups:
- Overall: Participants received JNJ-70033093 ( either 25 mg, 50 mg, 100 mg or 200 mg ) once daily or twice daily orally for 10 to 14 postoperative days.
Arm/Group | Overall
Number analyzed (Participants) | 921
Liter per hour (L/h) | 7.72 (39.5)

20. Secondary Outcome: Apparent Volume of Distribution (V/F) of JNJ-70033093
Description: V/F was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug.
Time Frame: Up to Day 14
Population: The PK analysis set consisted of participants who received at least 1 dose of milvexian and had at least one valid blood sample drawn for PK analysis. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure. This outcome measure was planned to be analyzed for overall participants and not group wise.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Overall
Number analyzed (Participants) | 921
Liter | 125 (60.5)

21. Secondary Outcome: Impact of Selected Demographics: Apparent Clearance (CL/F) Based on Sex
Description: Impact of demographic character (sex) on CL/F was assessed.
Time Frame: Up to Day 14
Population: The PK analysis set consisted of participants who received at least 1 dose of milvexian and had at least one valid blood sample drawn for PK analysis. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure. Arms are created based on sex (male and female) to report the effect of sex on CL/F.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/h)
Groups:
- Female: Participants received JNJ-70033093 ( either 25 mg, 50 mg, 100 mg or 200 mg) once daily or twice daily orally for 10 to 14 postoperative days.
- Male: Participants received JNJ-70033093 (either 25 mg, 50 mg, 100 mg or 200 mg) once daily or twice daily orally for 10 to 14 postoperative days.
Arm/Group | Female | Male
Number analyzed (Participants) | 653 | 268
Liter per hour (L/h) | 7.14 (38.5) | 9.32 (34.2)

22. Secondary Outcome: Impact of Selected Demographic: Age on CL/F
Description: Impact of age on CL/F was assessed.
Time Frame: Up to Day 14
Population: The PK analysis set consisted of participants who received at least 1 dose of milvexian and had at least one valid blood sample drawn for PK analysis. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure. Arms are created based on age to report the effect of age on CL/F.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Groups:
- Age: Less Than or Equal to (<=) 68 Years; Age: Greater Than (>) 68 Years: Participants received JNJ-70033093 (either 25 mg, 50 mg, 100 mg or 200 mg) once daily or twice daily orally for 10 to 14 postoperative days.
Arm/Group | Age: Less Than or Equal to (<=) 68 Years | Age: Greater Than (>) 68 Years
Number analyzed (Participants) | 464 | 457
L/h | 8.70 (36.9) | 6.83 (37.7)

23. Secondary Outcome: Impact of Selected Demographic: Weight on CL/F
Description: Impact of weight on CL/F was assessed.
Time Frame: Up to Day 14
Population: The PK analysis set consisted of participants who received at least 1 dose of milvexian and had at least one valid blood sample drawn for PK analysis. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure. Arms are created based on weight to report the effect of weight on CL/F.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Groups:
- Weight: <= 82 Kilograms (kg): Participants with weight <= 82 kg received an oral dose either of 25mg once daily, 50 mg once daily , 25mg BID, 50 mg BID, 200 mg once daily, 100 mg BID and enoxaparin once daily SC along with matching placebo for 10 to 14 postoperative days.
- Weight: Greater Than (>) 82 kg: Participants with weight > 82 kg received an oral dose either of 25mg once daily, 50 mg once daily , 25mg BID, 50 mg BID, 200 mg once daily, 100 mg BID and enoxaparin once daily SC along with matching placebo for 10 to 14 postoperative days.
Arm/Group | Weight: <= 82 Kilograms (kg) | Weight: Greater Than (>) 82 kg
Number analyzed (Participants) | 486 | 435
L/h | 7.04 (37.9) | 8.54 (38.4)

24. Secondary Outcome: Impact of Selected Laboratory Values: Renal Function on CL/F
Description: Impact of renal function on CL/F was assessed. The outcome measure was reported based on CRCL.
Time Frame: Up to Day 14
Population: The PK analysis set consisted of participants who received at least 1 dose of milvexian and had at least one valid blood sample drawn for PK analysis. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure. Arms are created based on CRCL to report the effect of renal function on CL/F.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Groups:
- Creatinine Clearance (CRCL): Less Than (<) 90; CRCL: Greater Than or Equal to (>=) 90: Participants received JNJ-70033093 (either 25 mg, 50 mg, 100 mg or 200 mg) once daily or twice daily orally for 10 to 14 postoperative days.
Arm/Group | Creatinine Clearance (CRCL): Less Than (<) 90 | CRCL: Greater Than or Equal to (>=) 90
Number analyzed (Participants) | 442 | 447
L/h | 6.71 (38.1) | 8.83 (35.1)

25. Secondary Outcome: Impact of Selected Demographics: Sex on Apparent Volume of Distribution (V/F)
Description: Impact of sex on V/F was assessed.
Time Frame: Up to Day 14
Population: The PK analysis set consisted of participants who received at least 1 dose of milvexian and had at least one valid blood sample drawn for PK analysis. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure. Arms are created based on sex (male and female) to report the effect of sex on V/F.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Groups:
- Female; Male: Participants received JNJ-70033093 (either 25 mg, 50 mg, 100 mg or 200 mg) once daily or twice daily orally for 10 to 14 postoperative days.
Arm/Group | Female | Male
Number analyzed (Participants) | 653 | 268
Liters | 118 (61.2) | 143 (56.0)

26. Secondary Outcome: Impact of Selected Demographics : Age on V/F
Description: Impact of age on V/F was assessed.
Time Frame: Up to Day 14
Population: The PK analysis set consisted of participants who received at least 1 dose of milvexian and had at least one valid blood sample drawn for PK analysis. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure. Arms are created based on age to report the effect of age on V/F.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Groups:
- AGE <= 68 Years: Participants aged <=68 years received an oral dose either of 25mg once daily, 50 mg once daily , 25mg BID, 50 mg BID, 200 mg once daily, 100 mg BID and enoxaparin once daily SC along with matching placebo for 10 to 14 postoperative days.
- AGE >68 Years: Participants received JNJ-70033093 (either 25 mg, 50 mg, 100 mg or 200 mg) once daily or twice daily orally for 10 to 14 postoperative days.
Arm/Group | AGE <= 68 Years | AGE >68 Years
Number analyzed (Participants) | 464 | 457
Liters | 135 (59.5) | 116 (60.3)

27. Secondary Outcome: Impact of Selected Demographics : Weight on V/F
Description: Impact of weight on V/F was assessed.
Time Frame: Up to Day 14
Population: The PK analysis set consisted of participants who received at least 1 dose of milvexian and had at least one valid blood sample drawn for PK analysis. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure. Arms are created based on weight to report the effect of weight on V/F.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Groups:
- Weight <= 82kg: Participants with weight <= 82 kg received an oral dose either of 25mg once daily, 50 mg once daily , 25mg BID, 50 mg BID, 200 mg once daily, 100 mg BID and enoxaparin once daily SC along with matching placebo for 10 to 14 postoperative days.
- Weight > 82kg: Participants with weight > 82 kg received an oral dose either of 25mg once daily, 50 mg once daily , 25mg BID, 50 mg BID, 200 mg once daily, 100 mg BID and enoxaparin once daily SC along with matching placebo for 10 to 14 postoperative days.
Arm/Group | Weight <= 82kg | Weight > 82kg
Number analyzed (Participants) | 486 | 435
Liters | 109 (58.8) | 145 (57.5)

28. Secondary Outcome: Impact of Selected Laboratory Values: Renal Function on V/F
Description: Impact of renal function on V/F was assessed. The outcome measure is reported based on CRCL.
Time Frame: Up to Day 14
Population: The PK analysis set consisted of participants who received at least 1 dose of milvexian and had at least one valid blood sample drawn for PK analysis. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure. Arms are created based on CRCL to report the effect of renal function on V/F.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Groups:
- CRCL < 90; CRCL >= 90: Participants received JNJ-70033093 (either 25 mg, 50 mg, 100 mg or 200 mg) once daily or twice daily orally for 10 to 14 postoperative days.
Arm/Group | CRCL < 90 | CRCL >= 90
Number analyzed (Participants) | 442 | 447
Liters | 116 (62.2) | 135 (58.5)

29. Secondary Outcome: Trend Test for Primary Efficacy Event Rate (CEC Adjudicated) by Multiple Comparison Procedure - Modelling (MCP-Mod) Approach
Description: The dose-response trend test based on the MCP-Mod framework consisted of contrast tests defined by prespecified candidate models (4 Emax dose-response models with varying degrees of ED50). Each model was evaluated for significance of trend, based on its optimal contrast, resulting in four t-test statistics, one for each candidate model. The t-test statistics were adjusted for the fact that 4 candidate models were included in the trend testing. The dose response of the drug was then established if the maximum of the t-test statistics exceeded the 95th percentile critical value. Here 'number' signifies the estimated response rate.
Time Frame: Up to 14 days
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | JNJ-70033093 25 mg Once Daily + Placebo | JNJ-70033093 50 mg Once Daily + Placebo | JNJ-70033093 25 mg + Placebo Twice Daily (BID) | JNJ-70033093 50 mg BID | JNJ-70033093 200 mg Once Daily + Placebo | JNJ-70033093 100 mg + Placebo BID | JNJ-70033093 200 mg BID
Number analyzed (Participants) | 28 | 127 | 129 | 124 | 123 | 134 | 131
proportion of participants | 0.35 [0.17 to 0.52] | 0.21 [0.16 to 0.25] | 0.20 [0.15 to 0.24] | 0.13 [0.10 to 0.16] | 0.09 [0.07 to 0.12] | 0.09 [0.06 to 0.11] | 0.07 [0.03 to 0.10]
Statistical Analysis 1: Comparison: JNJ-70033093 25 mg + Placebo Twice Daily (BID) vs JNJ-70033093 50 mg BID vs JNJ-70033093 100 mg + Placebo BID vs JNJ-70033093 200 mg BID; Test type: Other; p = 0.0004, MCP-mod analysis

30. Secondary Outcome: Trend Test for the Composite of On-Treatment Major and Clinically Relevant Nonmajor Bleeding (CEC Adjudicated) by MCP-Mod Approach
Description: as for outcome 29
Time Frame: Up to 14 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- JNJ-70033093 25 mg Once Daily + Placebo: Participants received JNJ-70033093 25 milligrams (mg) (1*25 mg capsule) once daily and 1 placebo capsule in the morning and 2 placebo capsules in the evening, orally for 10 to 14 postoperative.
  days.
Arm/Group | JNJ-70033093 25 mg Once Daily + Placebo | JNJ-70033093 50 mg Once Daily + Placebo | JNJ-70033093 25 mg + Placebo Twice Daily (BID) | JNJ-70033093 50 mg BID | JNJ-70033093 200 mg Once Daily + Placebo | JNJ-70033093 100 mg + Placebo BID | JNJ-70033093 200 mg BID
Number analyzed (Participants) | 33 | 150 | 148 | 148 | 147 | 149 | 148
proportion of participants | 0.02 [0.00 to 0.17] | 0.01 [0.00 to 0.03] | 0.01 [0.00 to 0.04] | 0.01 [0.00 to 0.02] | 0.01 [0.00 to 0.02] | 0.01 [0.00 to 0.02] | 0.01 [0.00 to 0.02]
Statistical Analysis 1: Comparison: JNJ-70033093 25 mg + Placebo Twice Daily (BID) vs JNJ-70033093 50 mg BID vs JNJ-70033093 100 mg + Placebo BID vs JNJ-70033093 200 mg BID; Test type: Other; p = 0.7188, MCP-MOD analysis

ADVERSE EVENTS:
Time Frame: Up to 6 weeks
Description: The safety analysis set is a subset of the intent to treat (ITT) analysis set, consisting of all ITT participants who received at least 1 dose (partial or complete) of study drug.
Arm/Group | JNJ-70033093 25 mg Once Daily + Placebo | JNJ-70033093 50 mg Once Daily + Placebo | JNJ-70033093 25 mg + Placebo Twice Daily (BID) | JNJ-70033093 50 mg BID | JNJ-70033093 200 mg Once Daily + Placebo | JNJ-70033093 100 mg + Placebo BID | JNJ-70033093 200 mg BID | Enoxaparin 40 mg Once Daily
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/150 | 0/148 | 0/148 | 0/147 | 0/149 | 0/148 | 1/296
Serious Adverse Events (participants affected / at risk) | 1/33 | 2/150 | 5/148 | 5/148 | 2/147 | 5/149 | 2/148 | 11/296
Other Adverse Events (participants affected / at risk) | 0/33 | 6/150 | 9/148 | 8/148 | 3/147 | 4/149 | 3/148 | 17/296
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | JNJ-70033093 25 mg Once Daily + Placebo (N=33) | JNJ-70033093 50 mg Once Daily + Placebo (N=150) | JNJ-70033093 25 mg + Placebo Twice Daily (BID) (N=148) | JNJ-70033093 50 mg BID (N=148) | JNJ-70033093 200 mg Once Daily + Placebo (N=147) | JNJ-70033093 100 mg + Placebo BID (N=149) | JNJ-70033093 200 mg BID (N=148) | Enoxaparin 40 mg Once Daily (N=296)
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device Related Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wound Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Periprosthetic Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiovascular Evaluation (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Full Blood Count Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin Decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Compartment Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ischaemic Stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 1 | 1 | 1 | 0 | 2 | 0 | 0
Femoral Artery Embolism (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | JNJ-70033093 25 mg Once Daily + Placebo (N=33) | JNJ-70033093 50 mg Once Daily + Placebo (N=150) | JNJ-70033093 25 mg + Placebo Twice Daily (BID) (N=148) | JNJ-70033093 50 mg BID (N=148) | JNJ-70033093 200 mg Once Daily + Placebo (N=147) | JNJ-70033093 100 mg + Placebo BID (N=149) | JNJ-70033093 200 mg BID (N=148) | Enoxaparin 40 mg Once Daily (N=296)
Constipation (Gastrointestinal disorders) | 0 | 6 | 9 | 8 | 3 | 4 | 3 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/24/NCT03891524/Prot_002.pdf
  • Statistical Analysis Plan (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/24/NCT03891524/SAP_003.pdf